CLINICAL TRIAL: NCT03697681
Title: Protective Effect of Tranexamic Acid on Shedding of the Endothelial Glycocalyx in Patients Undergoing Spinal Fusion Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4-2018-0754
Record Dates: First submitted 2018-10-01; First posted 2018-10-05 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Posterior Lumbar Spinal Fusion Surgery
MeSH Terms: interventions — Tranexamic Acid; Glutamine; Saline Solution

STUDY DESIGN:
Intervention Model Description: A Randomized, Double-Blinded, Placebo-Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: triple blinded (Participant, Care Provider, investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glutamine (Experimental): Intravenous glutamine infusion perioperatively for 18 hours (8 hours before surgery and 10 hours after induction of anesthesia)
  Interventions: Drug: Tranexamic acid
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: 0.9% NaCl (normal saline)

INTERVENTIONS:
Drug: Tranexamic acid — Intravenous infusion of Tranexamic acid(mixed with normal saline) at the dose of 10mg/kg(body weight) for 20 min after induction of anesthesia and then administration another 1mg/kg/hr(body weight) of Tranexamic acid(mixed with normal saline) until the end of the operation.
  Other Names: glutamine
  Arms: Glutamine
Drug: 0.9% NaCl (normal saline) — The same amount of normal saline solution without the addition of tranexamic acid is administered in the same manner as the experimental group(Tranexamic acid intervention group).
  Arms: Placebo

SUMMARY:
The aim of this study was to determine whether the administration of tranexamic acid in patients undergoing lumbar spinal fusion surgery can inhibit damage in endothelial glycocalyx layer. As a prospective double blinded randomized placebo-controlled trial, the investigators detect and compare the changes in concentrations of serum syndecan-1 and heparan sulfate before and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with between 30 and 80 years scheduled for posterior lumbar spinal fusion surgery.

Exclusion Criteria:

* emergency surgery
* patients unable to make their own decisions, illiterate, foreigners
* Allergy / hypersensitivity to Tranexamic acid
* Current or past history or thrombosis / thromboembolism
* patients who are taking oral contraceptives
* Patients with renal insufficiency (eGFR 60 ml / min / 1.73 m 2 or less)
* Patients receiving anticoagulants
* pregnant and lactating women

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2020-08-12 (Actual)

PRIMARY OUTCOMES:
base blood concentration of syndecan-1, heparan sulfate | within 1 hour before surgery(base concentration)
  preoperative baseline serum levels of syndecan-1 and heparan sulfate
blood concentration of syndecan-1, heparan sulfate at the end of the surgery | within 5 minutes after the end of surgery (when thd surgical drape is removed)
  blood concentration of syndecan-1, heparan sulfate at the end of the surgery
blood concentration of syndecan-1, heparan sulfate at 2 hours after surgery | 2 hours after the end of surgery
  blood concentration of syndecan-1, heparan sulfate at 2 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided